CLINICAL TRIAL: NCT03933111
Title: Application of Newly Developed Endoscopic Ultrasound With Zone Sonography Technology for Diagnosis of Pancreatic Caner: a Prospective Multicenter Study
Brief Title: Application of Newly Developed Endoscopic Ultrasound With Zone Sonography Technology for Diagnosis of Pancreatic Caner
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shengjing Hospital (Other); Beijing Friendship Hospital (Other); Huashan Hospital (Other); Sun Yat-sen University (Other); Tongji Hospital (Other); Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Department, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: shengsu
Record Dates: First submitted 2019-04-09; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Cancer
Keywords: Endoscopic Ultrasound; Zone Sonography Technology
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: All subjects are scanned by Fuji film su-9000 ultrasonic system. After the lesions are found, local sound velocity measurement technology will be used to measure the sound velocity in the lesions.Pathology diagnosis or clinical follow-up results will be regard as diagnostic gold standard to divide the patients into pancreatic cancer and pancreatic cancer group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with pancreatic solid neoplasms (Experimental): Patients with pancreatic solid neoplasms are enrolled in this study and accept the test.
  Interventions: Diagnostic Test: local sound velocity measurement

INTERVENTIONS:
Diagnostic Test: local sound velocity measurement — All patients are scanned by Fuji film su-9000 ultrasonic system. After the lesions are found, local sound velocity measurement technology will be used to measure the sound velocity in the lesions.Pathology diagnosis or clinical follow-up results will be regard as diagnostic gold standard divide the patients into pancreatic cancer and pancreatic cancer group.

SUMMARY:
The purpose of this study is to measure and compare the difference of sound speed between pancreatic cancer and non-pancreatic cancer, and determine the critical value of sound speed for benign and malignant pancreatic cancer. The sensitivity, specificity, accuracy, positive predictive value and negative predictive value for the diagnosis of pancreatic cancer are calculated, so as to evaluate the clinical application value of local sound speed measurement in the diagnosis of pancreatic cancer.

DETAILED DESCRIPTION:
The investigators include patients who are found to have solid pancreatic mass on continuous imaging. All subjects are scanned by Fuji film su-9000 ultrasonic system. After the lesions are found, local sound velocity measurement technology will be used to measure the sound velocity in the lesions. Pathology diagnosis or clinical follow-up results will be regard as diagnostic gold standard to divide the patients into pancreatic cancer and pancreatic cancer group. The investigators will compare the sound velocity value if there is statistically significant difference between the two groups, build the receiver operating characteristic curve, calculation of pancreatic benign and malignant lesions of sound velocity threshold, and and the investigators will calculate the sensitivity, specificity, accuracy, positive predictive value and negative predictive value, to evaluate local sound velocity measurement in the diagnosis of pancreatic cancer clinical application value.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 75, gender is not limited.
2. Evidence of solid pancreatic lesions have been found on imaging examination, including computed tomography, magnatic resonance imaging and endoscopic ultrasonography.
3. The lesion was greater 1cm.
4. The informed consent has been signed.

Exclusion Criteria:

1. Patients with serious cardiopulmonary diseases and poor general condition.
2. Patients with other contraindications to endoscopic ultrasonography.
3. Cannot or refuse to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
The threshold value of sound velocity for benign and malignant pancreatic lesions | up to 3 months
  The participants will compare the sound velocity value if there is statistically significant difference between the two groups, build the Receiver Operating Characteristic curve, determine the threshold value of sound velocity for benign and malignant pancreatic lesions.
The evaluation of the threshold value | up to 3 months
  The participants will calculate the sensitivity, specificity, accuracy, positive predictive value and negative predictive value, to evaluate local sound velocity measurement in the diagnosis of pancreatic cancer clinical application value.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-shen Li, M.D, Principal Investigator — Department of Gastroenterology, Changhai Hospital, Second Military Medical University
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No